CLINICAL TRIAL: NCT05572411
Title: Gait Analysis With Idiopathic Clubfoot Patients Treated by the Ponseti Method: Can Regular Assessment With the GAITRite Walkway Identify Common Gait Changes in Relapsing Patients?
Brief Title: Gait Analysis in Idiopathic Clubfoot Patients Treated by the Ponseti Method
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 13NS23
Record Dates: First submitted 2022-09-29; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Congenital Talipes Equino Varus
Keywords: CTEV; Clubfoot
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ponseti: Ponseti treated Clubfoot participants will be asked to walk across the GAITRite Electronic Walkway.
  Interventions: Other: GAITRite Electronic Walkway

INTERVENTIONS:
Other: GAITRite Electronic Walkway — Participants will be asked to walk across the electronic walkway to record information relating to their gait pattern. Depending on the age and compliance of the participant, they will be asked to complete 3 passes at 3 speeds, preferred, fast and slow.

SUMMARY:
The purpose of this study is to assess the walking pattern of clubfoot patients using a pressure sensing walkway, and investigate whether any of the data produced can be used to detect the early signs of relapse in their foot posture.

DETAILED DESCRIPTION:
Study Background:

A series of studies have used the GAITRite Electronic Walkway to collect normative data with more than 500 typically developing children between the ages of 1 - 18 years of age. The data was used to produce novel normative gait related percentile charts. These charts provide an immediate reference against which individual scores can be plotted and improvements demonstrated. Their value in the clinical setting was demonstrated by the inclusion of a variety of clinical diagnoses which all have the ability to affect the gait pattern. One clinical group consisted of Ponseti treated Idiopathic Clubfoot patients.

Gait is an important functional milestone for all children, particularly if the child has undergone treatment to produce a functional foot position which will allow them to engage in normal childhood activities with minimal pain and discomfort. Treatment concepts in Clubfoot are centred on non-operative techniques where the outcome is improved by avoiding the scar tissue associated with surgical releases. Gait analysis results at medium and long term intervals support the improved functional ability following non-operative intervention however infrequent analysis has resulted in a lack of longitudinal gait analysis in the Clubfoot population. Such information would give an insight into the development of gait in the presence of a corrected deformity being challenged by the rapid growth of the child.

The gait analysis systems used in many of the published research are complex, expensive and require specialised skills to operate, presenting many barriers to performing regular gait analysis. In contrast, the GAITRite is a relatively inexpensive, portable, child friendly system which allows for frequent gait analysis, producing Temporo-spatial data, easily extracted and interpreted by the clinician. From the longitudinal data we would be able to study the development of gait and pressure patterns within this patient population, investigating whether particular parameters or trends exist that are indicative of relapse in foot posture, aiding early identification and implementation of treatment.

Aims and Objectives:

The aim of this research project is to incorporate gait analysis with the GAITRite electronic walkway into the assessment of patients attending the GOSH Ponseti clinic. This will provide on-going information regarding the development of gait and response of the deformity correction to growth in these patients.

The objective is to analyse the data and determine if it is possible to identify common clinical measures which will help determine patients at greater risk of relapse.

Practical Details:

Ambulant patients who have received Ponseti treatment for Idiopathic CTEV will be identified through the GOSH Ponseti clinic and invited to participate in the study.

As part of their assessment at each appointment, height, weight and leg length data will be measured and the participants will be asked to walk across the 6m pressure sensing walkway. Depending on the age of the child and ability to follow instruction, the participant will be asked to walk at self-selected, fast and slow speed, with 4 repetitions at each one. The participant will start walking 2m before the walkway and continue 2m after it, to allow for recording of a steady gait. The process takes approximately 15 minutes per child.

Data Collection/Storage:

The personal data required for each participant is their name and date of birth. These will be collected in paper form on the consent and screening form, after which the participant will be assigned a study number and be referred to as such in collecting and storing electronic data. All manual forms will be securely stored in a locked cabinet on Trust premises in line with the Trust policy for storing patient records.

With regards to the electronic data, as previously stated, participants will be identified by number rather than name. The Gaitrite data initially be stored on a laptop but will be uploaded as soon as possible to the Trust server and the laptop data being removed by the appropriate means. Access to the Gaitrite and Trust server is via log in and individual password.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Congenital Talipes Equinovarus
* Received Ponseti method for management of their deformity.
* Ambulant

Exclusion Criteria:

* Syndromic Clubfoot

Ages: 12 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of Idiopathic Congenital Talipes Equinovarus patients who received the Ponseti Method for management of their deformity.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Gait Related Relapse Indicator | Bi-annually for duration of follow-up at GOSH between 2-7 years
  Assessment in clinic GAITRite electronic walkway is able to identify specific gait parameters which suggest deterioration in the correction achieved with the initial Ponseti management, these will be presented as a way of combining clinical assessment with instrumented gait analysis for thorough evaluation of the patients progress.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kemp, Bsc (Hons), Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Result] Eastwood, D., Alderson, LM, Kemp J. Measuring consistency of gait performance over 3 speeds with Ponseti Treated Club foot patients. J Child Orthopaedics. 2015. (S12) 9 Suppl1: S11-S5
- [Result] EPOS 34th Annual Meeting. J Child Orthop. 2015 Apr;9(Suppl 1):11-56. doi: 10.1007/s11832-015-0637-0. No abstract available. PMID 25754189